CLINICAL TRIAL: NCT07032194
Title: Use of the Da Vinci Single Port Robotic System in Urological Surgery: A Prospective Observational Study (SP-URO)
Brief Title: Prospective Study on the Use of the Da Vinci SP System in Urological Surgery
Acronym: SP-URO
Status: Recruiting | Type: Observational
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: 001-FPO25
Record Dates: First submitted 2025-05-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Urologic Surgical Procedure
Keywords: Da Vinci Single Port (SP) System; Urologic Surgery; multiport

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Da Vinci SP Robotic Surgery Cohort: This cohort includes all patients undergoing urologic surgical procedures using the Da Vinci Single Port (SP) robotic platform at IRCCS Candiolo. The procedures may include radical prostatectomy, partial or radical nephrectomy, adenomectomy, and nephroureterectomy. All surgeries are performed through a single surgical incision using the SP system, without additional experimental interventions. The outcomes of this cohort will be observed prospectively, and perioperative, functional, and oncologic results will be analyzed. Exploratory comparisons may be made with outcomes from historical or contemporaneous multiport (Da Vinci Xi) procedures

SUMMARY:
A prospective observational study aimed at evaluating the feasibility, safety, and effectiveness of the Da Vinci SP robotic system for urologic procedures at IRCCS Candiolo. The study collects perioperative, oncologic, and functional outcomes, with exploratory comparisons to the multiport Da Vinci Xi system.

DETAILED DESCRIPTION:
Minimally invasive surgery has significantly evolved with the introduction of robotic systems. The Da Vinci Single Port (SP) system, FDA-approved in 2018, allows procedures to be performed through a single incision. This single-center, prospective observational study conducted at IRCCS Candiolo aims to assess the safety, feasibility, and perioperative, oncologic, and functional outcomes of urologic procedures performed with the Da Vinci SP system.

Patients will be followed for up to 60 months post-surgery, with exploratory analysis comparing outcomes to those from procedures performed with the Da Vinci Xi (multiport) system. Data will include perioperative variables, complications, renal function, urinary continence, sexual potency, and oncologic parameters. Statistical analyses will be performed using Stata.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and data privacy consent
* Clinical indication for urologic robotic surgery per EAU guidelines or clinical trial eligibility
* ECOG Performance Status 0-1
* Life expectancy ≥ 10 years
* Availability of preoperative clinical data
* Willingness to comply with follow-up visits and data collection
* Eligibility for robotic surgery

Exclusion Criteria:

* Unsuitability for anesthesia
* Cognitive or psychiatric disorders affecting consent or compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age Range: 18 years and older Sex: All Healthy Volunteers: Not accepted Sampling Method: Non-probability sample Study Location: IRCCS Candiolo, Italy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Perioperative complication rate | Within 30 days post-surgery
  The complication rate will be evaluated using the Clavien-Dindo classification, tracking complications during the perioperative period (30 days after surgery).
Conversion rate of SP robotic surgery | Surgery through 30 postoperative days
  Feasibility of performing urologic surgeries using the Da Vinci SP system will be evaluated in terms of conversion rate to multiport surgeries or open approach

SECONDARY OUTCOMES:
Surgical margins | Up to 60 months
  Oncologic outcomes will include:
  - the evaluation of surgical margins (occurrence of positive surgical margin - PSM at final pathology examination)
BCR | Up to 60 months
  Oncologic outcomes will include:
  - biochemical recurrence rates (BCR- defined as presence of biochemical recurrence for prostate cancer as PSA > 0.2 ng/dl; or presence of new tumoral lesions or metastasis for kidney and urothelial cancer)
CSM | Up to 60 months
  Oncologic outcomes will include:
  - long-term survival for patients who underwent oncologic urologic surgery.in terms of cancer specific mortality (CSM)
OM | Up to 60 months
  Oncologic outcomes will include:
  - overall mortality (OM)
Continence recovery | 3 to 60 months post-surgery
  This outcome will track urinary continence post-surgery, assessing the impact of the robotic approach on patients' quality of life.
  Continence will be defined as "total continence" (o pads) o "social continence" (1 safety pad).
Potency | 3 to 60 months post-surgery
  This outcome will track sexual potency post-surgery, assessing the impact of the robotic approach on patients' quality of life.
  Potency will be defined as erection sufficient for intercourse or masturbation. IPSS and IEEF-5 questionnaires will be administered during the follow-up.
Renal Function | 3 to 60 months post-surgery
  This outcome will trackrenal function post-surgery, assessing the impact of the robotic approach on patients' quality of life.
  It will be evaluated in terms of eGFR drop
Exploratory Endpoints (Comparison to Da Vinci Xi System) | End-of-study analysis (60 months)
  An exploratory analysis will compare the Da Vinci SP system to the Da Vinci Xi multiport system.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione del Piemonte per l'Oncologia- IRCCS Istituto di Candiolo, Candiolo, Turin, Italy

IPD SHARING:
Plan to Share IPD: No